CLINICAL TRIAL: NCT04743115
Title: A Phase I, Open-Label, Dose Escalation and Cohort Expansion Study of BS HH 002.SA in Patients With Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: A Phase I, Open-Label, Dose Escalation and Cohort Expansion Study of BS HH 002.SA in Patients With AML and MDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Bensen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BS HH 002.SA
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia, Myelodysplastic Syndrome
Keywords: BS HH 002.SA
MeSH Terms: conditions — GATA2 Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- the Dose Escalation Level (Experimental): In the first 3-patient cohort, the dose of BS HH 002.SA will be 0.2 mg/m2/day. Enrollment to the next higher dose cohort will be initiated only if none of the 3 patients exhibits a DLT in the first 28-day cycle. Dose escalation will proceed according to a modified Fibonacci scheme, eg, increments of 100%, 100%, 66%, and 33% and the dose of BS-HH-002.SA will be 0.4, 0.8, 1.3, 1.7 mg/m2/day.
  The dose will be administered subcutaneously once daily on Days 1 through 6 and on Days 10 through 15 of a 28 day cycle.
  Interventions: Drug: BS HH 002.SA

INTERVENTIONS:
Drug: BS HH 002.SA — The Dose Escalation Part is a 3+3 design dose escalation study to determine the MTD of BS HH 002.SA in up to approximately 30 patients with the protocol AML indication or high risk MDS. Cohorts of 3 patients will be sequentially assigned to receive BS HH 002.SA at escalating DLs following the standard 3+3 dose escalation design, with 3 to 6 patients at each DL.
  Cohort Expansion Part: Following determination of the MTD, the study will continue at the MTD and/or a lower DL

SUMMARY:
Indication:Relapsed or refractory AML in patients for whom no established treatment options are available (this indication will heretofore be referred to as the protocol AML indication), or adult patients with MDS who are classified as high risk or very high risk according to the Revised International Prognosis Scoring System (IPSS-R).

Number of Investigators and Study Centers:Up to 5 Investigators in the US. Objectives:Dose Escalation Part

Primary Objective:

1. To determine the maximum tolerated dose (MTD) of BS HH 002.SA administered subcutaneously once per day for 12 days of a 28-day cycle.

   Secondary Objectives:
2. To provide an initial safety profile of single and multiple cycles of BS HH 002.SA.
3. To assess the pharmacokinetic (PK) profile of BS HH 002.SA.
4. To explore the anti-tumor activity of BS HH 002.SA in patients with the protocol AML indication or high-risk MDS.
5. To explore cytogenetics of the malignant cells in relation to response to BS HH 002.SA.

Cohort Expansion Part

Primary Objectives:

1. To evaluate safety and tolerability of BS HH 002.SA at MTD and/or lower dose level (DL) in selected cohorts of patients with the protocol AML indication or high-risk MDS.
2. To evaluate preliminary anti-tumor activity of BS HH 002.SA at MTD and/or lower DL in selected cohorts of patients with the protocol AML indication or high-risk MDS.

   Secondary Objectives:
3. To assess the PK profile of BS HH 002.SA.
4. To explore cytogenetics of the malignant cells in relation to response to BS HH 002.SA.

Study Population:Adult patients with the protocol AML indication or high-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥18 years of age
2. Patients with one of the following conditions:

   1. Primary or secondary AML, pathologically confirmed according to World Health Organization (WHO) or IWG classification, who have relapsed or refractory disease and for whom no established treatment options are available, or who are not a candidate for current therapies
   2. High risk or very high risk MDS, as evaluated according to the IPSS R, who are resistant or intolerant to standard treatment and not candidates for transplantation
3. Patients must be willing to participate in the study and have the ability to understand and adhere to study visit schedule and other protocol procedures. They should be able to comprehend and willing to sign an Informed Consent Form (ICF)
4. Women of childbearing potential must have two negative pregnancy tests during Screening, the second within 24 hours prior to the first administration of study drug, and must agree to use highly effective physician-approved contraception from Screening to 90 days following the last study drug administration. For the purposes of this study, women with tubal ligations are considered to be of childbearing potential but women who are surgically sterile (hysterectomy) or post menopausal ≥2 years are not considered to be of childbearing potential Note: Post-menopausal is defined as aged more than 50 years and amenorrhea for at least 12 months following cessation of all exogenous hormonal treatment. Women with irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation, are acceptable.
5. Male subjects must be surgically sterile. If male subjects are able to father children, they must use a highly effective physician-approved birth control method from Screening, during the study, and for 90 days after the last dose of study drug. The study physician will inform the subject which birth control methods are acceptable. Vasectomy and sexual abstinence are the recommended birth control methods Note: Female partners of male subjects should not become pregnant during the course of the study as the effects of the study drug on an unborn child and on a breast-fed baby are not known. Male participants will not be allowed to take part in this study if their female partner is trying to become pregnant. If female partner does become pregnant while male partner is taking part in the study, male participants should immediately inform the study physician. The female partner will be asked to sign a Pregnant Partner Data Release Form.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status 3 or greater
2. Known hypersensitivity to study drug or its excipients
3. Acute promyelocytic leukemia
4. Administration of any antineoplastic therapy or anti-MDS treatment within at least 2 weeks or 5 half-lives (whichever is greater) of the first dose of BS HH 002.SA, with the exception of hydroxyurea for AML patients which should be discontinued 1 day prior to the first dose of BS HH 002.SA
5. Participation in other clinical trials within at least 2 weeks of the first BS HH 002.SA dose
6. Concomitantly receiving other investigational agents
7. Clinical evidence of active central nervous system leukemia
8. History of diabetes mellitus and a hemoglobin A1c ≥7.0% as assessed at Screening
9. Active and uncontrolled infection including but not limited to known infection with HIV, active hepatitis B, or hepatitis C. Patients with an infection receiving treatment with antibiotics may be entered into the trial if they are afebrile and hemodynamically stable for 96 hours prior to trial entry
10. Major surgery within 2 weeks prior to trial entry
11. Receipt of an allogeneic or autologous stem cell transplant within 60 days of the first BS HH 002.SA dose
12. Toxicities from a previous anti-cancer therapy that are NCI CTCAE Grade 2 or greater, except for alopecia and Grade 2 nausea
13. Liver function tests above the following limits at Screening: total bilirubin >1.5 × upper limit of normal (ULN) unless related to Gilbert's syndrome or hemolysis, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 × ULN, or for patients with liver involvement AST and/or ALT >5 × ULN
14. Liver malignancy (including metastases) or chronic liver disease
15. Previous drug-induced liver injury (DILI)
16. Serum creatinine >1.5 × ULN and/or creatinine clearance (CrCl) <30 mL/min at Screening (calculation according to Cockcroft & Gault formula or Modification of Diet in Renal Disease [MDRD] formula)
17. International normalized ratio (INR) >1.5 × ULN, or, if on warfarin therapy, INR >2.5 × ULN
18. Corrected QT interval (QTc) by Fridericia's method (QTcF) >450 msec or concomitant use of drugs known to prolong the QTc (antiemetic therapy can be allowed with approval from the Medical Monitor if the QTc is normal, and calcium, magnesium, and potassium levels are normal on Day 1)
19. New York Heart Association class III or IV heart disease, uncontrolled hypertension, congestive heart failure, or other uncontrolled cardiac condition
20. Left ventricular ejection fraction (LVEF) <45% as assessed by multiple-gated acquisition (MUGA) scan or echocardiogram
21. Uncontrolled congestive heart failure, unstable angina pectoris
22. Patients with concomitant solid tumors or lymphoma, for whom the Investigator has clinical suspicion of active disease at the time of enrolment. Patients with adequately treated early-stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia, or with castrate sensitive prostate cancer with stable elevated prostate-specific antigen under anti-androgenic therapy are eligible for this study
23. Other significant disease that in the Investigator's opinion would exclude the patient from the participation in the study protocol
24. Women who are or plan to become pregnant, or who are currently breastfeeding
25. Active alcohol or drug abuse
26. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Part: the maximum tolerated dose (MTD) of BS HH 002.SA administered subcutaneously once per day for 12 days of a 28-day cycle. | the first 28 day cycle
Cohort Expansion Part: To evaluate safety and tolerability of BS HH 002.SA at MTD and/or lower dose level (DL) in selected cohorts of patients with the protocol AML indication or high-risk MDStreatment | maximum of 12 months
Cohort Expansion Part: To evaluate preliminary anti-tumor activity of BS HH 002.SA at MTD and/or lower DL in selected cohorts of patients with the protocol AML indication or high-risk MDS. | maximum of 12 months

IPD SHARING:
Plan to Share IPD: No